CLINICAL TRIAL: NCT02006537
Title: A Study to Evaluate the Effect of Age, Food and Gender on Tolerability and Pharmacokinetics of GSK2256294 Following a Single Oral Administration in Healthy Fed and Fasted Elderly Subjects. This Study Will Also Evaluate the Biliary Metabolites in Healthy Young Males Following a Single Dose of GSK2256294
Brief Title: A Study to Investigate the Safety and Pharmacokinetics of a Single Dose of GSK2256294 in Healthy Young Males and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117023
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: soluble epoxide hydrolase inhibitor; Entero-Test; pharmacokinetics; COPD; safety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N-((4-cyano-2-(trifluoromethyl)phenyl)methyl)-3-((4-methyl-6-(methylamino)-1,3,5-triazin-2-yl)amino)cyclohexanecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will enrol 8 healthy male volunteers, who will receive a single 10 mg dose of GSK225694 in the fasted state.
  Interventions: Drug: GSK2256294
- Cohort 2 (Experimental): Cohort 2 will enrol 20 healthy elderly male and female volunteers (10 males and 10 females), who will receive a single 10 mg dose of GSK225694 in the fasted or fed state according to the randomization schedule.
  Interventions: Drug: GSK2256294

INTERVENTIONS:
Drug: GSK2256294 — GSK2256294 is a 5 mg capsule administered orally as a 10 mg dose in the fasted or fed state

SUMMARY:
This study will investigate the safety and pharmacokinetics (PK) of a single dose of GSK2256294 in healthy young and elderly subjects to explore the effects of food, gender and age on drug exposure. The biliary metabolites in healthy young males will be investigated using the Entero-test after a single oral dose of GSK2256294. This study will be conducted in two cohorts (Cohort 1 and Cohort 2). Cohort 1 is open label in order to characterise the PK profile of GSK2256294 in healthy young males and also to investigate the biliary metabolites of GSK2256294. Cohort 2 uses a crossover design to allow comparison of the PK parameters of GSK2256294 between in the fed and fasted state within subject and also to compare the PK parameters of GSK2256294 between male and female subjects. A washout period of a minimum of 2 weeks has been chosen to allow and adequate washout of GSK2256294.

ELIGIBILITY:
Inclusion Criteria:

* Safety - All Cohorts
* 12 lead ECG without any clinically significant abnormality as judged by the Investigator, and ECGs QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 milliseconds (msec) determined by the average of triplicate ECGs.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 2 weeks post-last dose.
* Body weight >=60 kilogram (kg) and body mass index (BMI) within the range 19 - 35 kg per meter square (kg/m^2) (inclusive).
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5xUpper limit of normal [ULN] (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter outside the reference range for the population being studies may be included only of the Investigator agree that the finding is unlikely to introduce additional risk factors and will not interfere with study procedures. Consultation with the GSK Medical Monitor is required.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Safety - Cohort 2 Only
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international units per milliliter (mIU/mL) and estradiol <40 picogram per milliliter (pg/mL) (<147 picomole per liter) is confirmatory]. [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods listed in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]
* Other - Cohort 1 Only.
* Cohort 1 only: Male aged between 18 and 45 years of age inclusive, at the time of signing the informed consent.

Cohort 1 only: BP <=130/80.

* Other - Cohort 2 Only
* Cohort 2 only: Male and females (of non-child bearing potential) aged >=60 years of age, at the time of signing the informed consent.
* Cohort 2 only: BP <=160/100.

Exclusion Criteria:

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).

* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for human immunodeficiency virus (HIV) antibody.
* A positive pre-study drug/alcohol screen.
* Subjects with a history of any type of malignancy with the exception of successfully treated squamous cell cancer of the skin.
* History of sensitivity to the study medication, or components thereof or a history of drug allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicated their participation.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2014-05-27 (Actual); Study Completion 2014-05-27 (Actual)

PRIMARY OUTCOMES:
Cohort 2: PK profiles of a single oral dose of GSK2256294 | Pre-dose, 15 minutes (min), 30 min, 1 hour (h), 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h (Day 1) and 24 h (Day 2), 48 h (Day 3) and 72 h (Day 4)
  PK parameters including area under the concentration-time curve (AUC) and maximum blood concentrations (Cmax), half life (T1/2), time to Cmax (Tmax) following a single oral dose of GSK2256294 administered under fed and fasted conditions in healthy elderly male and female subjects will be estimated
Cohort 2: Electrocardiogram (ECG) as a measure of safety and tolerability | Screening, Pre-dose, 30 min, 2 h, 4 h, 6 h and at follow-up
  Twelve-lead ECGs will be obtained as a measure of safety and tolerability
Cohort 2: Adverse events (AEs ) as a measure of safety and tolerability | From the start of study treatment and until approximately 2 weeks after the final dose
Cohort 2: Vital signs as a measure of safety and tolerability | Screening, Pre-dose, 30 min, 2 h, 4 h, 6 h and at follow-up
  Vital sign measurements will include systolic and diastolic blood pressure (BP) and pulse rate
Cohort 2: Laboratory assessments as a measure of safety and tolerability | Screening and follow-up. In addition, clinical chemistry will also be done at 12 h (Day 1) and 24 h (Day 2)
  Clinical laboratory assessments will include haematology, clinical chemistry, urinalysis and other screening tests

SECONDARY OUTCOMES:
Cohort 1: Biliary metabolite profile of GSK2256294 | Until 7 hours post-dose on Day 1
  Bile will be collected for metabolic analysis of GSK2256294 + metabolites via the use of the Entero-Test capsule in healthy male younger subjects
Cohort 1: AEs as a measure of safety and tolerability | From the start of study treatment and until approximately 2 weeks after the final dose
Cohort 1: ECG as a measure of safety and tolerability | Screening, Pre-dose, 30 min, 2 h, 4 h, 6 h and at follow-up
  Twelve-lead ECGs will be obtained to assess safety and tolerability
Cohort 1: Vital signs as a measure of safety and tolerability | Screening, Pre-dose, 30 min, 2 h, 4 h, 6 h and at follow-up
  Vital sign measurements will include systolic and diastolic BP and pulse rate
Cohort 1: Laboratory assessments as a measure of safety and tolerability | Screening and follow-up
  Clinical laboratory assessments will include haematology, clinical chemistry, urinalysis and other screening tests
Cohort 1 and Cohort 2: AUC, Cmax, t1/2,and Tmax of GSK2256294 | Cohort 1: Pre-dose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 7 h, 12 h and 24 h, 48 h, and 72 h; Cohort 2: Pre-dose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h and 24 h, 48 h and 72 h
  To compare the pharmacokinetic profiles of single oral doses of GSK2256294 in healthy elderly and healthy younger subjects, and between healthy elderly male and female subjects

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lazaar AL, Yang L, Boardley RL, Goyal NS, Robertson J, Baldwin SJ, Newby DE, Wilkinson IB, Tal-Singer R, Mayer RJ, Cheriyan J. Pharmacokinetics, pharmacodynamics and adverse event profile of GSK2256294, a novel soluble epoxide hydrolase inhibitor. Br J Clin Pharmacol. 2016 May;81(5):971-9. doi: 10.1111/bcp.12855. Epub 2016 Jan 17. PMID 26620151
- See also: Results for study 117023 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117023?search=study&search_terms=117023#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 117023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register